CLINICAL TRIAL: NCT06859034
Title: Therapeutic Effect of Proliferative Therapy (prolotherapy) on Pain Using Injectable Hypertonic Dextrose 25% Versus Injectable Dextrose 10% in Retrodiscal Tissues in Patients with Anterior Disc Displacement with Reduction: a Randomized Clinical Trial .
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Moustafa, dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: prolotherapy injection in tmj
Record Dates: First submitted 2025-02-22; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: TMJ Disc Disorder
Keywords: retrodiscal tissues

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- injection of dextrose 10% in retrodiscal tissues (Active Comparator): GROUP 1 will recieve 10% dextrose
  Interventions: Drug: injection of dextrose 10% in retrodiscal tissues
- injection of dextrose 25% in retrodiscal tissues (Experimental): group 2 will recieve 25% dextrose
  Interventions: Drug: injection of dextrose 25% in retrodiscal tissues

INTERVENTIONS:
Drug: injection of dextrose 10% in retrodiscal tissues — group 1 will recieve 10% dextrose in retrodiscal tissues
  Arms: injection of dextrose 10% in retrodiscal tissues
Drug: injection of dextrose 25% in retrodiscal tissues — group 2 will recieve 25% dextrose
  Arms: injection of dextrose 25% in retrodiscal tissues

SUMMARY:
prolotherapy is an injection-based treatment method used to alleviate pain, particularly musculoskeletal pain associated with chronic ligament and tendon injuries. The process involves the injection of a solution, typically containing dextrose (a sugar), saline, or other irritants, into the affected tissues. Prolotherapy is believed to stimulate healing by causing a mild inflammatory response that promotes the regeneration of ligaments, tendons, and other connective tissues. This review explores the existing literature on the therapeutic effects of prolotherapy for pain management.

DETAILED DESCRIPTION:
Anterior disc displacement with reduction (ADDR) is a common temporomandibular joint (TMJ) disorder, characterized by the displacement of the articular disc in front of the condyle during mouth opening, which then reduces upon closing. This condition often results in pain, restricted jaw movement, and clicking sounds. Conservative treatments, including physical therapy, splint therapy, and pharmacological interventions, are commonly used, but these may not always yield long-term results. Recent studies have explored the role of prolotherapy, particularly the use of dextrose injections, in treating TMJ disorders, including ADDR. Among the variations in prolotherapy, the concentration of dextrose solution-commonly 10% and 25%-is often debated for its potential effectiveness in promoting healing and pain relief. Prolotherapy is often compared to other injection-based treatments, such as corticosteroid injections and platelet-rich plasma (PRP) therapy. A study by Chou et al. (2017) found that prolotherapy was more effective than corticosteroid injections for the management of chronic tendon and ligament pain, with longer-lasting effects and fewer side effects. Similarly, prolotherapy was found to be as effective as PRP for certain conditions, such as chronic tendinopathies, although PRP may offer additional benefits in tissue regeneration due to its higher concentration of growth factors (Gosens et al., 2020).

6

The literature supports prolotherapy as a promising treatment for various chronic pain conditions, especially those involving tendons, ligaments, and joints. Evidence from clinical trials suggests that prolotherapy is effective in reducing pain, improving function, and promoting tissue regeneration in conditions like chronic low back pain, knee osteoarthritis, and soft tissue injuries. However, despite the promising results, the overall quality of evidence remains moderate, and further large-scale, high-quality studies are needed to fully establish its efficacy and long-term outcomes. Prolotherapy is generally safe, but like any invasive treatment, it carries a risk of adverse effects, albeit minimal.

As prolotherapy continues to gain recognition in pain management, its potential as an adjunct or alternative to traditional therapies warrants further investigation.

ELIGIBILITY:
Exclusion criteria:

* The clinical or radiographic signs of disc displacement without reduction .
* A history of allergic reactions to any components of the injectable solution.
* Blood dyscrasias and systemtic diseases .
* Previous surgery of the affected joint.
* Infection in pre-auricular area

Inclusion criteria:

Patients should have one or more signs and symptoms of these

* Symptoms: Patients who report typical symptoms of TMJ dysfunction, such as pain, discomfort, or clicking sounds in the joint, especially when opening or closing the mouth.
* Mouth Opening: Limited range of motion or difficulty with full mouth opening .
* Clicking: Audible clicking.
* Pain: Pain or tenderness around the TMJ, often radiating to the ear, temple, or neck

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2025-09-03 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Severity Measured by Numerical Rating Scale (NRS) | Measured at baseline, 1 month, 3 months, and 6 months after injections.
  Pain severity will be assessed using the Numerical Rating Scale (NRS) (0-10), where 0 = no pain and 10 = severe pain. Participants will report their pain levels at each time point. The mean change in NRS scores from baseline will be calculated and analyzed . Data Aggregation: Mean change in NRS score with standard deviation (SD)

SECONDARY OUTCOMES:
Change in Maximal Interincisal Opening (MIO) Measured in Millimeters | Measured at baseline, 1 month, 3 months, and 6 months after injections
  Maximal interincisal opening (MIO) will be measured using a digital caliper, with values recorded in millimeters (mm). The mean change in MIO from baseline will be reported . Data Aggregation: Mean change in MIO (mm) with standard deviation (SD).
Presence or Absence of Joint Clicking (Binary Outcome) | Measured at baseline, 1 month, 3 months, and 6 months after injections
  Joint clicking will be assessed as a binary outcome (Yes/No) based on clinical examination and patient-reported symptoms. The percentage of participants with joint clicking at each time point will be reported.
  Data Aggregation: Percentage of participants with joint clicking at each time point

CONTACTS AND LOCATIONS:
Overall Officials: nadia galal Professor, phd, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Haggag MA, Al-Belasy FA, Said Ahmed WM. Dextrose prolotherapy for pain and dysfunction of the TMJ reducible disc displacement: A randomized, double-blind clinical study. J Craniomaxillofac Surg. 2022 May;50(5):426-431. doi: 10.1016/j.jcms.2022.02.009. Epub 2022 Mar 8. PMID 35501215
- [Background] Park JS, Ku JK, Kim YK, Yun PY. Efficacy of dextrose prolotherapy on temporomandibular disorder: a retrospective study. J Korean Assoc Oral Maxillofac Surg. 2024 Oct 31;50(5):259-264. doi: 10.5125/jkaoms.2024.50.5.259. PMID 39482101